CLINICAL TRIAL: NCT04318080
Title: A Phase 2, Multicenter, Open-Label Study of Tislelizumab (BGB-A317) in Patients With Relapsed or Refractory Classical Hodgkin Lymphoma
Brief Title: Tislelizumab in Participants With Relapsed or Refractory Classical Hodgkin Lymphoma
Acronym: TIRHOL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Collaborators: Lymphoma Study Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-210; 2019-002105-22 (EudraCT Number)
Record Dates: First submitted 2020-03-20; First posted 2020-03-23 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Classical Hodgkin Lymphoma
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Participants who had relapsed or refractory classical Hodgkin lymphoma and had either not achieved a response or had disease progression following autologous hematopoietic stem cell transplantation received tislelizumab 200 milligrams (mg) intravenously every 3 weeks.
  Interventions: Drug: Tislelizumab
- Cohort 2 (Experimental): Participants who had relapsed or refractory classical Hodgkin lymphoma and had either not achieved a response or had disease progression after at least one prior systemic therapy and were not candidates for autologous or allogeneic hematopoietic stem cell transplantation received tislelizumab 200 mg intravenously every 3 weeks.
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — 200 milligrams (mg) intravenously every 3 weeks (Q3W)
  Other Names: BGB-A317

SUMMARY:
This was a Phase 2 trial evaluating the effectiveness and safety of tislelizumab in participants with relapsed or hard-to-treat classical Hodgkin lymphoma (cHL). Participants were grouped by prior treatments. The main outcome was to assess overall response rate (ORR) across both cohorts. Participants continued receiving the study treatment until their disease got worse, side effects became too severe, or they chose to stop for other reasons.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants had a histologically confirmed diagnosis of relapsed or refractory classical Hodgkin lymphoma (cHL).
2. Participants had either:

   * Relapsed cHL, defined as disease progression after a partial response (PR) or complete response (CR) to their most recent therapy; or
   * Refractory cHL, defined as failure to achieve PR or CR to their most recent therapy.

   Participants were assigned to one of two cohorts based on the following:

   Cohort 1: Participants who were relapsed or refractory after prior autologous hematopoietic stem cell transplantation (HSCT):
   1. Had failed to achieve a response or had experienced disease progression following autologous HSCT (a transplant using the participant's own stem cells).
   2. Were not considered candidates for additional autologous or allogeneic HSCT (a transplant using donor stem cells).

   Cohort 2: Participants who were relapsed or refractory to salvage chemotherapy and had not received prior HSCT:
   1. Were not considered candidates for autologous or allogeneic HSCT.
   2. Had received at least one prior systemic therapy regimen for cHL.
3. Participants had measurable disease, defined as at least one positron emission tomography (PET)-positive, 2-\[18F] fluoro-2-deoxy-D-glucose (FDG)-avid nodal lesion greater than 1.5 centimeters (cm) in longest diameter, or at least one FDG-avid extranodal lesion (hepatic nodule) greater than 1.0 cm in longest diameter.
4. Participants had an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1, indicating full activity or restricted activity but capable of self-care.

Key Exclusion Criteria:

1. Participants had nodular lymphocyte-predominant Hodgkin lymphoma or gray zone lymphoma.
2. Participants had received prior allogeneic HSCT.
3. Participants had received prior therapy targeting immune checkpoint pathways, including programmed cell death protein 1 (PD-1), programmed death-ligand 1 (PD-L1), programmed death-ligand 2 (PD-L2), or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4).
4. Participants had active autoimmune disease or a history of autoimmune disease with potential to relapse.

Note: Additional inclusion and exclusion criteria defined in the protocol may have applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2024-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herve Ghesguieres, Principal Investigator — Lymphoma Study Association
Locations (4):
- United States (3):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Monash Health, Clayton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved. BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations. Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/

REFERENCES:
- [Result] Ghesquières H, López-Guillermo A, De la Cruz F, et al. Tislelizumab, an anti-PD-1 antibody, in patients with relapsed/refractory classical Hodgkin lymphoma in TIRHOL BGB-A317-210: a prospective multicenter LYSA phase 2 study conducted in Western countries. Blood. 2023;142(Suppl 1):1717. DOI:10.1182/blood-2023-188545
- [Result] Ghesquières H, et al. TIRHOL (BGB-A317-210): International Phase 2 Study in Relapsed/Refractory Classical Hodgkin Lymphoma. Presented at: Congrès de la Société Française d'Hématologie (SFH); March 2024; Paris, France.
- [Result] Ghesquières H, López-Guillermo A, De la Cruz F, et al. Final analysis from the LYSA phase 2 TIRHOL study (BGB-A317-210): tislelizumab in relapsed/refractory classical Hodgkin lymphoma. Presented at: 18th International Conference on Malignant Lymphoma (ICML); June 18-22, 2025; Lugano, Switzerland. https://doi.org/10.1002/hon.70093_130

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at multiple centers across France, the United States, Belgium, and Australia from August 20, 2020, to August 29, 2024.
Pre-assignment Details: After enrollment, open-label tislelizumab treatment began. Screening was completed within 28 days before the first dose. Treatment started within 14 days of eligibility confirmation, within the screening window. Treatment continued until disease progression, unacceptable toxicity, or withdrawal. Participants who did not meet eligibility criteria during screening were excluded prior to assignment to treatment groups.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 15 | 31
Treated | 14 | 31
Completed | 0 | 0
Not Completed | 15 | 31
Not completed — Study closed by sponsor | 10 | 22
Not completed — Death | 3 | 9
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Deviation | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 14 | 31 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.9 (15.78) | 59.6 (21.95) | 54.7 (21.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 11 | 15
  Male | 10 | 20 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 5 | 8
  Not Reported | 11 | 26 | 37
Patient Status at Time of Enrollment [Count of Participants; unit: Participants] — Refractory refers to participants whose disease did not respond to their most recent prior therapy (no complete or partial response). Relapse/Progression refers to participants whose disease initially responded to prior therapy but later worsened, progressed, or returned.
  Participants
    Refractory | 0 | 13 | 13
    Relapse/Progression | 14 | 18 | 32
The Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) Performance Status is a standard scale used to assess how a participant's disease impacts their daily living abilities. It ranges from 0 (fully active) to 5 (dead), with higher scores indicating greater functional impairment.
  Participants
    0 (Normal activities) | 10 | 18 | 28
    1 (Ambulatory able to carry out work) | 4 | 13 | 17
Number of prior lines of therapy for cHL [Count of Participants; unit: Participants]
  1 | 0 | 7 | 7
  2 | 9 | 17 | 26
  3 | 4 | 6 | 10
  4 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved a best overall response of complete response (CR) or partial response (PR) by Positron Emission Tomography (PET) and Computed Tomography (CT) per the Lugano Classification and as determined by the investigator. CR was defined as the complete disappearance of all target lesions on PET-CT, with no new lesions detected. PR was defined as a significant reduction in metabolic activity or lesion size consistent with partial tumor shrinkage as per Lugano criteria.
Time Frame: From first dose to primary analysis data cutoff (12 Dec 2022) or new anti-lymphoma therapy start, whichever came first. Median follow-up was 11.4 months.
Population: Safety Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Total: Participants received tislelizumab 200 mg intravenously every 3 weeks.
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 14 | 31 | 45
Percentage of Participants | 64.3 [35.1 to 87.2] | 64.5 [45.4 to 80.8] | 64.4 [48.8 to 78.1]
Statistical Analysis 1: Comparison: Total; The primary analysis was conducted on both cohorts combined, A binomial exact test was performed to test the null hypothesis (H0: ORR = 45% based on previous clinical trials) and alternative hypothesis (ORR >45%). If the one-sided p-value was ≤ 0.05, tislelizumab was considered to statistically significantly increase ORR compared to the historical control; Test type: Superiority — Analysis tested whether ORR with tislelizumab was superior to a historical ORR of 45% using a one-sided binomial exact test (α = 0.05); p = 0.0044, Binomial Exact Test — One-sided p-value based on a binomial exact test comparing observed ORR to historical rate of 45%; Z-test = 2.62

2. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR was defined as the percentage of participants who achieved a best overall response of complete response (CR) by PET-CT or CT per the Lugano Classification and determined by the investigator. CR was defined as the complete disappearance of all target lesions on PET-CT or CT, with no new lesions detected.
Time Frame: as for outcome 1
Population: Safety Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 14 | 31 | 45
Percentage of Participants | 42.9 [17.7 to 71.1] | 25.8 [11.9 to 44.6] | 31.1 [18.2 to 46.6]

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the date that response criteria (CR or PR) were first met to the date of objectively documented disease progression or death, whichever occurred first. Participants without an event were censored at the data cutoff or end of study, whichever occurred first. Participants who received new anti-lymphoma therapies, including Hematopoietic Stem Cell Transplantation (HSCT), before having an event were censored at the date of therapy initiation. Only participants with confirmed response were included in the analysis. Median DOR was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: The responder analysis set only included participants with a confirmed response (CR) or partial response (PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 9 | 20 | 29
months | 12.25 [5.55 to 12.25] | 6.64 [2.79 to NA] — Not estimable due to insufficient number of participants with events | 12.25 [3.02 to NA] — Not estimable due to insufficient number of participants with events

4. Secondary Outcome: Time to Response (TTR)
Description: TRR was defined as the time from the date of the first dose of tislelizumab to the date the response criteria were first met CR or PR per the Lugano Classification, and was analyzed only in participants who achieved an overall response; CR was defined as complete disappearance of disease, PR as ≥50% reduction in tumor burden, and Overall Response Rate (ORR) included participants with either CR or PR.
Time Frame: as for outcome 1
Population: Safety Analysis Set. Only participants who had achieved an overall response were included in the analysis of time to response.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 9 | 20 | 29
months | 2.69 [2.1 to 5.5] | 2.69 [0.3 to 5.6] | 2.69 [0.3 to 5.6]

5. Secondary Outcome: Number of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Adverse events (AEs) were assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0. Treatment-emergent adverse events (TEAEs) were defined as any AE that began or worsened in severity after the first dose of study treatment and up to 90 days following the last dose, regardless of initiation of new anti-lymphoma therapy. The following safety data are reported:
  Number of participants with any TEAEs: Participants who experienced at least one TEAE of any grade.
  Number of participants with any Grade ≥3 TEAEs: Participants who experienced at least one TEAE that was Grade 3 or higher in severity.
  Number of participants with any SAEs: Participants who experienced at least one serious adverse event, regardless of relationship to study treatment, occurring up to 90 days after the last dose.
Time Frame: From the date of the first dose of tislelizumab through 90 days after the last dose (maximum duration of tislelizumab exposure was 168 weeks)
Population: Safety Analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 14 | 31
Participants
  Number of participants with any TEAEs | 12 | 30
  Number of participants with any TEAEs with grade >= 3 | 4 | 12
  Number of participants with any SAEs | 4 | 9

ADVERSE EVENTS:
Time Frame: All-cause mortality was reported from randomization to 29 Aug 2024 (4 years). AEs were reported from first tislelizumab dose to 90 days post-last dose (max exposure: 168 weeks).
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 3/14 | 9/31
Serious Adverse Events (participants affected / at risk) | 4/14 | 9/31
Other Adverse Events (participants affected / at risk) | 12/14 | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=14) | Cohort 2 (N=31)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cutaneous t-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=14) | Cohort 2 (N=31)
Anaemia (Blood and lymphatic system disorders) | 1 (5) | 4 (4)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 0 (0) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1)
Hyperadrenocorticism (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1) | 4 (4)
Chalazion (Eye disorders) | 0 (0) | 1 (1)
Periorbital swelling (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 4 (4)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (6)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 3 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Asthenia (General disorders) | 1 (2) | 9 (16)
Chest pain (General disorders) | 0 (0) | 3 (3)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 4 (6)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 3 (4) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (4)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 1 (1)
Balanoposthitis infective (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (3) | 3 (3)
COVID-19 (Infections and infestations) | 1 (1) | 3 (3)
Conjunctivitis (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Dermo-hypodermitis (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0)
Oral infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 2 (3)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (6)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (14) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Steroid diabetes (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (3)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 4 (4)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1)
Bulimia nervosa (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus urethral (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT04318080/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT04318080/SAP_001.pdf